CLINICAL TRIAL: NCT05684107
Title: Femoral Nerve Block Combined With Sciatic Nerve Block Adductor Canal Block Or (Interspace Between The Popliteal Artery And The Capsule Of The Posterior Knee) IPACK Block For Postoperative Analgesia After Major Knee Surgeries
Brief Title: Sciatic Nerve Block, Adductor Canal Block, or IPACK Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, mostafa saieed fahim mansour, lecturer, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 10/2022ANETH2
Record Dates: First submitted 2022-12-20; First posted 2023-01-13 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Post Operative Pain
Keywords: IPACK , Sciatic nerve block , adductor canal block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IPACK block (Active Comparator)
  Interventions: Procedure: IPACK block
- sciatic nerve block (Active Comparator)
  Interventions: Procedure: sciatic nerve block
- adductor canal block (Active Comparator)
  Interventions: Procedure: adductor canal block

INTERVENTIONS:
Procedure: IPACK block — the probe is applied to the popliteal fossa for identification of the popliteal artery and femur. Then, the probe is slid distally for revealing the two femoral condyles followed by proximal sliding of the probe until the humps of the femoral condyles disappeared and the flat metaphysis appeared. a spinal needle 22G x 3.5 inches is advanced from the lateral aspect and directed across the space between the popliteal artery and femur and once the needle reached the medial edge of the femur, nearly at the level of the popliteal artery, negative aspiration is confirmed and 20 ml of bupivacaine 0.25% is injected incrementally as the needle was withdrawn
  Arms: IPACK block
Procedure: adductor canal block — the transducer is placed anteromedially, approximately at the junction between the middle and distal third of the thigh or somewhat lower.
  The saphenous nerve block should be performed at the most distal level where the artery still lies immediately deep to the sartorius muscle, thus minimizing the amount of motor nerve block of the vastus medialis; an adductor canal nerve block is typically performed more proximally, around the mid-thigh level. The needle is inserted in-plane in a lateral-to-medial orientation and advanced toward the femoral artery. Once the needle tip is visualized anterior to the artery and after careful aspiration, 20 ml of bupivacaine 0.25% is injected incrementally as the needle was withdrawn
  Arms: adductor canal block
Procedure: sciatic nerve block — patient in a supine position with the hip and knee on the operated side flexed and the leg externally rotated at approximately 45 degrees. The ultrasound transducer is first positioned perpendicular to the skin approximately 8 cm distal to the inguinal crease. The location is then scanned by sliding and tilting the transducer until a clear transverse image of the hyperechoic sciatic nerve located posterior and medial to the lesser trochanter is obtained. a spinal needle 22G x 3.5 inches is advanced parallel and in line with the ultrasound transducer while the sciatic nerve is kept in the middle of the screen. The needle is advanced slowly under real-time ultrasound guidance until it is near the nerve then negative aspiration is confirmed and 20 ml of bupivacaine 0.25% is injected incrementally as the needle was withdrawn
  Arms: sciatic nerve block

SUMMARY:
Comparison between local anesthetic infiltration between the popliteal artery and the capsule of the knee (IPACK) versus adductor canal block (ACB) or sciatic nerve block (anterior approach) in combination with femoral nerve block for postoperative analgesia in major knee surgeries.

ELIGIBILITY:
Inclusion Criteria:

* ASA I or II physical status
* undergoing elective major knee surgery

Exclusion Criteria:

* refusal of the patients to give informed consent,
* preexisting coagulation disorders,
* known allergies to aminoamide local anesthetics,
* local infection at the site of the block,
* morbid obesity,
* hepatic and renal diseases
* patients with psychological disorders

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
change of visual analogue scale | change from 0 level every 1 hour for 1st 6 hours,then every 4 hours for next 24 hours and on movement
  a scale from 0 to 10 as the patient will be asked to express his pain on the scale higher scale means a worse outcome

SECONDARY OUTCOMES:
time for fisrt analgesic request | up to 48 hours
  when VAS is 4 or more longer time means a better outcome
total morphine consumption | up to 48 hours
  intraoperative and post operative higher consumption means a worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, University Hospitals, Shibīn al Kawm, Menoufia, Egypt